CLINICAL TRIAL: NCT05272215
Title: Longitudinal Follow-up and Comparison of Bariatric and Post-bariatric Body Contouring Patient's Health-related Quality of Life Relative to Population Norms Using the BODY-Q
Brief Title: BODY-Q Longitudinal Result Study and Comparison With Normative Scores
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Hospital of Southwest Jutland, Esbjerg, Denmark (Unknown); McMaster University (Other); OLVG West Hospital, Amsterdam, the Netherlands (Unknown); Catharina Ziekenhuis Eindhoven (Other); Tampere University Hospital (Other); Department of Plastic Surgery, Wroclaw, Poland (Unknown); Department of Plastic Surgery, Eberhard Karls Universität Tübingen, Tübingen, Germany (Other); Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Farima Dalaei, MD, Odense University Hospital
Other Study IDs: 10240356
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Weight Loss; Excess Skin
Keywords: Bariatric surgery; Massive weight loss; Body contouring surgery; Health-related quality of life; Quality of life; Post bariatric surgery
MeSH Terms: conditions — Weight Loss | interventions — Bariatric Surgery; Body Contouring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient group: Pre-BaS: Patients administered for BaS, Department of Endocrinology either Odense University Hospital, Odense, Denmark or Hospital of Southwest Jutland, Esbjerg, Denmark
  Post-BaS: (3, 6, 12 months postoperatively, then yearly) Department of Surgery, Southwest Jutland, Esbjerg, Denmark
  Pre-BC: Patients administered for BC, Department of Plastic Surgery, Odense University Hospital, Odense, Denmark or Department of Plastic Surgery, Southwest Jutland, Esbjerg, Denmark.
  Post-BC: (3, 6, 12 months postoperatively, then yearly), department of Plastic Surgery, Odense University Hospital; Hospital of Southwest Jutland, Esbjerg.
  Normative group: Reference scores of the general population from an international sample of 10 countries and country specific scores. This study sample is submitted for publication elsewhere.
  Interventions: Procedure: Bariatric surgery; Procedure: Body contouring surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Pre- and post-bariatric surgery (3, 6, 12 months postoperative and yearly)
Procedure: Body contouring surgery — Pre- and post body contouring surgery (3, 6, 12 months postoperative and yearly)

SUMMARY:
Obesity is a global epidemic that has nearly tripled since 1975. Worldwide, over 650 million people live with obesity, and it is therefore a growing cause for concern. Bariatric surgery (BaS) is the most effective long-term weight loss method in morbidly obese patients. BaS can result in sustained weight loss and resolve obesity-related comorbidities. However, BaS most often results in various extremes of excess skin, where subsequent body contouring surgery (BC) can be needed. The excess skin following massive weight loss is known to negatively impacts patients' body image, physical and psychological well-being, which previous studies have indicated to improve after BC.

The purpose of this study is to assess change in patients' health-related quality of life (HRQL) relative to the general population score. To the best of our knowledge, there are no studies measuring change of patient's HRQL throughout the entire weight loss journey and comparing these scores with the scores of the general population.

It is hypothesized that 1) BaS will improve patients' quality of life on short terms (1-2 years) after surgery, however patients' HRQL will decrease with increasing amounts of excess skin. 2) Patients' HRQL will improve after post-BC equivalent of the scores of the general population.

DETAILED DESCRIPTION:
HRQL is best measured through patient-reported outcomes (PRO), defined as a patient evaluation of outcomes without interference from clinicians or any other intermediary. A vast array of patient-reported outcome measure (PROM)s have been used in weight loss and BC patients, many of which do not possess strong evidence of reliability and validity for the patient population.

In 2016, The BODY-Q, a condition-specific PROM developed following internationally recommended guidelines to measure PRO in weight loss, including bariatric surgery, and body contouring surgery (BC) patients were introduced. It consists of 32 independently functioning scales measuring four domains: appearance, HRQL, eating-related concerns, and patient experience of care. It is rigorously tested to ensure content validity, reliability, and responsiveness. Due to the strongest evidence for validity and its psychometric properties, recent systematic review based on the Consensus-based Standards for the selection of health Measurement Instruments (COSMIN) methodology only recommend the BODY-Q for use in this patient population.

The BODY-Q has been shown to be responsive to change and subsequently to measure change over the entire weight loss trajectory, i.e., from obesity to weight loss with or without BC. In previous studies, the BODY-Q has been used to demonstrate the efficacy of weight loss therapy and BC.

However, a current limitation of the BODY-Q is the lack of general population norms as a reference value of the four domains (HRQL, appearance, eating-related concerns, and experience of care). To date, it is not known how published preoperative and postoperative scores compare to population norms, enabling a better understanding of HRQL of obesity and change through the weight loss trajectory.

The primary aim of this study is to investigate the change of HRQL through the entire weight loss journey from obesity to post-BC in a longitudinal, prospective cohort study of Danish patients. The study will be performed as part of an international collaboration and Danish data will be merged with data from the Netherlands, Finland, Poland, Italy, Germany, and the United States. The secondary aim of this study is to compare international patient results with the general population norms. The general population norms. Currently, the general population norms study is under submission.

ELIGIBILITY:
Inclusion Criteria:

* Pre- and post-bariatric surgery patients
* Pre- and post body contouring surgery patients
* Fluent in Danish

Exclusion Criteria:

* Patients who do not speak Danish
* Patients with cognitive impairments
* Patients who have not undergone BaS/BC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Danish patients are recruited from June 2015 to May 2022 from four hospital departments in the Region of Southern Denmark: Department of Endocrinology, Hospital of Southwest Jutland; Department of Endocrinology, Odense University Hospital; Department of Plastic Surgery, Hospital of Southwest Jutland; and Department of Plastic Surgery, Odense University Hospital. Patients are asked to fill out the BODY-Q at following time points: before BaS, after BaS (3- ,6- ,12-months postoperative, then yearly) before BC, and after BC (3-, 6-, 12-months postoperative, then yearly). Data is collected using REDCap (Research Electronic Data Capture). The REDCap survey link and written information about the study were sent via patients' electronic secure mailbox.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
BODY-Q Health-related quality of life (HRQL) domain | June 2015 to May 2022
  Following scales are included:
  1. Appearance distress
  2. Body image
  3. Physical function
  4. Physical symptoms
  5. Psychological
  6. Sexual
  7. Social
  8. Work life

SECONDARY OUTCOMES:
Comparison of patient scores to general population normative scores | June 2015 to May 2022
  The scores of patients will be compared to the general population normative scores to assess the impact of BaS and BC on patients' lives compared to the general population HRQL.

CONTACTS AND LOCATIONS:
Overall Officials: Jens A Sørensen, MD, PhD, Principal Investigator — Odense University Hospital; Lotte Poulsen, MD, PhD, Principal Investigator — Odense University Hospital; Farima Dalaei, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Plastic Surgery, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan available for IPD sharing